CLINICAL TRIAL: NCT01822015
Title: A Pilot, Pharmacodynamic Correlate Trial of Sirolimus in Combination With Chemotherapy (Idarubicin, Cytarabine) for the Treatment of Newly Diagnosed Acute Myelogenous Leukemia
Brief Title: Sirolimus, Idarubicin, and Cytarabine in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12D.588; 2012-55 (Other: CCRRC); JT 3038 (Other: JeffTrial Number)
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Sirolimus; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (sirolimus, idarubicin, cytarabine) (Experimental): Patients receive sirolimus PO QD on days 1-10, idarubicin IV over 3-5 minutes on days 4-6, and cytarabine IV continuously over 24 hours on days 4-10.
  Interventions: Drug: Sirolimus; Drug: Idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: Sirolimus — Given PO
  Other Names: rapamycin; Rapamune
Drug: Idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; Zavedos; Idamycin
Drug: Cytarabine — Given IV
  Other Names: cytosine arabinoside; Cytosar-U; Depocyt; Ara-C; Arabinofuranosyl Cytidine

SUMMARY:
This pilot clinical trial studies sirolimus, idarubicin, and cytarabine in treating patients with newly diagnosed acute myeloid leukemia. Sirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving sirolimus together with idarubicin and cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1) To determine whether there is an association between baseline mammalian target of rapamycin (mTOR) activation paired with mTOR target inhibition post-treatment in leukemic blasts and clinical response in patients with newly diagnosed acute myeloid leukemia (AML) treated with sirolimus idarubicin/cytarabine.

SECONDARY OBJECTIVES:

1. To estimate the response rate of sirolimus idarubicin/cytarabine in patients with newly diagnosed AML compared to historical data using idarubicin/cytarabine alone.
2. To determine the ability of oral sirolimus to inhibit mTOR in leukemic blasts.
3. To assess if mTOR pathway inhibition correlates with clinical response.
4. To collect further information on the safety, tolerability, and efficacy of sirolimus in combination with idarubicin/cytarabine in patients with newly diagnosed AML.
5. To describe the progression-free survival and overall survival (1 year, 2 year and 5 year) of patients treated with sirolimus idarubicin/cytarabine.

OUTLINE:

Patients receive sirolimus orally (PO) once daily (QD) on days 1-10, idarubicin intravenously (IV) over 3-5 minutes on days 4-6, and cytarabine IV continuously over 24 hours on days 4-10.

After completion of study treatment, patients are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic evidence of newly diagnosed acute myeloid leukemia (non-M3 AML) as documented by the presence of >20% myeloid blasts in the bone marrow
2. Subjects must be 18 years of age and <= 60
3. Subjects must have an ECOG performance status of 2 or less. (see attachment 1).
4. Subjects must have a life expectancy of at least 4 weeks.
5. Subjects must be able to consume oral medication.
6. Required initial laboratory values: Creatinine 2.0mg/dL; total or direct bilirubin 1.5mg/dL; SGPT(ALT) 3xULN (if not due to the leukemia itself); negative pregnancy test for women with child-bearing potential.
7. Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
8. Subjects must have a left ventricular ejection fraction (LVEF) of >/= 45%.

Exclusion Criteria:

1. Subjects with APL - FAB M3 (t(15;17)(q22;q21)[PML-RAR] are not eligible
2. Subjects must not have received any chemotherapeutic agents for the AML (except Hydroxyurea). Intrathecal ARA-C and intrathecal methotrexate are permissible (as they are not systemic and only isolated to the central nervous system).
3. Subjects must not be receiving growth factors, except for erythropoietin.
4. Subjects with a "currently active" second malignancy, other than non-melanoma skin cancers are not eligible.
5. Subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, myocardial infarction within the past 6 months or serious uncontrolled cardiac arrhythmia are not eligible.
6. Subjects taking the following are not eligible:

   1. Carbamazepine (e.g., Tegretol)
   2. Rifabutin (e.g., Mycobutin)
   3. Rifampin (e.g., Rifadin)
   4. Rifapentine (e.g., Priftin)
   5. St. John's wort
   6. Clarithromycin (e.g., Biaxin)
   7. Cyclosporine (e.g. Neoral or Sandimmune)
   8. Diltiazem (e.g., Cardizem)
   9. Erythromycin (e.g., Akne-Mycin, Ery-Tab)
   10. Itraconazole (e.g., Sporanox)
   11. Ketoconazole (e.g., Nizoral)
   12. Telithromycin (e.g., Ketek)
   13. Verapamil (e.g., Calan SR, Isoptin, Verelan)
   14. Voriconazole (e.g., VFEND)
   15. Tacrolimus (e.g. Prograf)
7. Subjects taking fluconazole, voriconazole, itraconazole, posaconazole, and ketoconazole within 72 hours of study entry are not eligible. Reinstitution of fluconazole, voriconazole, itraconazole, posaconazole, ketoconazole and diltiazem is permissible 72 hours after the last dose of sirolimus.
8. Subjects who require HIV protease inhibitors or those with AIDS-related illness
9. Subjects with other severe concurrent disease which in the judgment of the investigator would make the patient inappropriate for entry into this study are ineligible.
10. Subjects must not be pregnant or breastfeeding. Pregnancy tests must be obtained for all females of child-bearing potential. Pregnant or lactating patients are ineligible for this study due to the unknown human fetal or teratogenic toxicities of sirolimus. Males or females of reproductive age may not participate unless they have agreed to use an effective contraceptive method.
11. Subjects who have uncontrolled infection are not eligible. Patients must have any active infections under control. Fungal disease must be stable for at least 2 weeks before study entry.
12. Subjects with bacteremia must have documented negative blood cultures prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Change in measurement of mTOR activation paired with mTOR target inhibition | Baseline to day 4
  The association between mTOR response and clinical response (complete or partial response) will be evaluated using the two-sided Fisher's exact test with alpha 0.05.

SECONDARY OUTCOMES:
Overall survival | 1 year, 2 years, 5 years
  Will be evaluated using the Kaplan-Meier method stratified by mTOR response. Log rank test will be used to compare the overall survival in patients with and without mTOR response. Based on the estimated survival curves, the 1-year, 2-year, and 5-year survival rates will be computed with the corresponding 95% confidence intervals.
Progression free survival | 1 year, 2 years, 5 years
  Based on the estimated survival curves, the 1-year, 2-year, and 5-year survival rates will be computed with the corresponding 95% confidence intervals.
Incidence of toxicities, graded according to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) 4.0 guidelines | Up to 45 days
  Safety data analysis is descriptive. All estimates of adverse events rates will be presented with corresponding confidence intervals using the exact method.
Response defined as patients achieving a complete remission (CR), complete response in absence of total platelet recovery (CRp), or partial remission (PR) | Up to 5 years
  Proportions of complete response and partial response with be computed separately in patients with and without mTOR response and presented with corresponding exact binomial 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kasner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bishop JF, Matthews JP, Young GA, Szer J, Gillett A, Joshua D, Bradstock K, Enno A, Wolf MM, Fox R, Cobcroft R, Herrmann R, Van Der Weyden M, Lowenthal RM, Page F, Garson OM, Juneja S. A randomized study of high-dose cytarabine in induction in acute myeloid leukemia. Blood. 1996 Mar 1;87(5):1710-7. PMID 8634416
- [Background] Gilliland DG, Jordan CT, Felix CA. The molecular basis of leukemia. Hematology Am Soc Hematol Educ Program. 2004:80-97. doi: 10.1182/asheducation-2004.1.80. PMID 15561678
- [Background] Castaigne S, Chevret S, Archimbaud E, Fenaux P, Bordessoule D, Tilly H, de Revel T, Simon M, Dupriez B, Renoux M, Janvier M, Miclea JM, Thomas X, Bastard C, Preudhomme C, Bauters F, Degos L, Dombret H. Randomized comparison of double induction and timed-sequential induction to a "3 + 7" induction in adults with AML: long-term analysis of the Acute Leukemia French Association (ALFA) 9000 study. Blood. 2004 Oct 15;104(8):2467-74. doi: 10.1182/blood-2003-10-3561. Epub 2004 May 13. PMID 15142880
- [Background] Stone RM. The difficult problem of acute myeloid leukemia in the older adult. CA Cancer J Clin. 2002 Nov-Dec;52(6):363-71. doi: 10.3322/canjclin.52.6.363. PMID 12469764
- [Background] Burnett AK, Hills RK, Milligan DW, Goldstone AH, Prentice AG, McMullin MF, Duncombe A, Gibson B, Wheatley K. Attempts to optimize induction and consolidation treatment in acute myeloid leukemia: results of the MRC AML12 trial. J Clin Oncol. 2010 Feb 1;28(4):586-95. doi: 10.1200/JCO.2009.22.9088. Epub 2009 Dec 28. PMID 20038732
- [Background] Buchner T, Berdel WE, Haferlach C, Haferlach T, Schnittger S, Muller-Tidow C, Braess J, Spiekermann K, Kienast J, Staib P, Gruneisen A, Kern W, Reichle A, Maschmeyer G, Aul C, Lengfelder E, Sauerland MC, Heinecke A, Wormann B, Hiddemann W. Age-related risk profile and chemotherapy dose response in acute myeloid leukemia: a study by the German Acute Myeloid Leukemia Cooperative Group. J Clin Oncol. 2009 Jan 1;27(1):61-9. doi: 10.1200/JCO.2007.15.4245. Epub 2008 Dec 1. PMID 19047294
- [Background] Cassileth PA, Harrington DP, Appelbaum FR, Lazarus HM, Rowe JM, Paietta E, Willman C, Hurd DD, Bennett JM, Blume KG, Head DR, Wiernik PH. Chemotherapy compared with autologous or allogeneic bone marrow transplantation in the management of acute myeloid leukemia in first remission. N Engl J Med. 1998 Dec 3;339(23):1649-56. doi: 10.1056/NEJM199812033392301. PMID 9834301
- [Background] Estey E. Acute myeloid leukemia and myelodysplastic syndromes in older patients. J Clin Oncol. 2007 May 10;25(14):1908-15. doi: 10.1200/JCO.2006.10.2731. PMID 17488990
- [Background] Mayer RJ, Davis RB, Schiffer CA, Berg DT, Sarno E, Frei E 3rd. Intensive post-remission therapy with Ara-C in adults with acute myeloid leukemia: initial results of a CALGB phase III trial. The Cancer and Leukemia Group B. Leukemia. 1992;6 Suppl 2:66-7. No abstract available. PMID 1578945
- [Background] Menzin J, Lang K, Earle CC, Kerney D, Mallick R. The outcomes and costs of acute myeloid leukemia among the elderly. Arch Intern Med. 2002 Jul 22;162(14):1597-603. doi: 10.1001/archinte.162.14.1597. PMID 12123403
- [Background] Bennett JM, Andersen JW, Cassileth PA. Long term survival in acute myeloid leukemia: the Eastern Cooperative Oncology Group (ECOG) experience. Leuk Res. 1991;15(4):223-7. doi: 10.1016/0145-2126(91)90124-c. PMID 2030603
- [Background] Weick JK, Kopecky KJ, Appelbaum FR, Head DR, Kingsbury LL, Balcerzak SP, Bickers JN, Hynes HE, Welborn JL, Simon SR, Grever M. A randomized investigation of high-dose versus standard-dose cytosine arabinoside with daunorubicin in patients with previously untreated acute myeloid leukemia: a Southwest Oncology Group study. Blood. 1996 Oct 15;88(8):2841-51. PMID 8874180
- [Background] Ohtake S, Miyawaki S, Fujita H, Kiyoi H, Shinagawa K, Usui N, Okumura H, Miyamura K, Nakaseko C, Miyazaki Y, Fujieda A, Nagai T, Yamane T, Taniwaki M, Takahashi M, Yagasaki F, Kimura Y, Asou N, Sakamaki H, Handa H, Honda S, Ohnishi K, Naoe T, Ohno R. Randomized study of induction therapy comparing standard-dose idarubicin with high-dose daunorubicin in adult patients with previously untreated acute myeloid leukemia: the JALSG AML201 Study. Blood. 2011 Feb 24;117(8):2358-65. doi: 10.1182/blood-2010-03-273243. Epub 2010 Aug 6. PMID 20693429
- [Background] Druker BJ, Talpaz M, Resta DJ, Peng B, Buchdunger E, Ford JM, Lydon NB, Kantarjian H, Capdeville R, Ohno-Jones S, Sawyers CL. Efficacy and safety of a specific inhibitor of the BCR-ABL tyrosine kinase in chronic myeloid leukemia. N Engl J Med. 2001 Apr 5;344(14):1031-7. doi: 10.1056/NEJM200104053441401. PMID 11287972
- [Background] Thomas DA, Faderl S, Cortes J, O'Brien S, Giles FJ, Kornblau SM, Garcia-Manero G, Keating MJ, Andreeff M, Jeha S, Beran M, Verstovsek S, Pierce S, Letvak L, Salvado A, Champlin R, Talpaz M, Kantarjian H. Treatment of Philadelphia chromosome-positive acute lymphocytic leukemia with hyper-CVAD and imatinib mesylate. Blood. 2004 Jun 15;103(12):4396-407. doi: 10.1182/blood-2003-08-2958. Epub 2003 Oct 9. PMID 14551133
- [Background] Thompson JE, Thompson CB. Putting the rap on Akt. J Clin Oncol. 2004 Oct 15;22(20):4217-26. doi: 10.1200/JCO.2004.01.103. PMID 15483033
- [Background] Bardet V, Tamburini J, Ifrah N, Dreyfus F, Mayeux P, Bouscary D, Lacombe C. Single cell analysis of phosphoinositide 3-kinase/Akt and ERK activation in acute myeloid leukemia by flow cytometry. Haematologica. 2006 Jun;91(6):757-64. PMID 16769577
- [Background] Xu Q, Simpson SE, Scialla TJ, Bagg A, Carroll M. Survival of acute myeloid leukemia cells requires PI3 kinase activation. Blood. 2003 Aug 1;102(3):972-80. doi: 10.1182/blood-2002-11-3429. Epub 2003 Apr 17. PMID 12702506
- [Background] Zhao S, Konopleva M, Cabreira-Hansen M, Xie Z, Hu W, Milella M, Estrov Z, Mills GB, Andreeff M. Inhibition of phosphatidylinositol 3-kinase dephosphorylates BAD and promotes apoptosis in myeloid leukemias. Leukemia. 2004 Feb;18(2):267-75. doi: 10.1038/sj.leu.2403220. PMID 14628071
- [Background] Edinger AL, Thompson CB. Akt maintains cell size and survival by increasing mTOR-dependent nutrient uptake. Mol Biol Cell. 2002 Jul;13(7):2276-88. doi: 10.1091/mbc.01-12-0584. PMID 12134068
- [Background] Wullschleger S, Loewith R, Hall MN. TOR signaling in growth and metabolism. Cell. 2006 Feb 10;124(3):471-84. doi: 10.1016/j.cell.2006.01.016. PMID 16469695
- [Background] Harada H, Andersen JS, Mann M, Terada N, Korsmeyer SJ. p70S6 kinase signals cell survival as well as growth, inactivating the pro-apoptotic molecule BAD. Proc Natl Acad Sci U S A. 2001 Aug 14;98(17):9666-70. doi: 10.1073/pnas.171301998. Epub 2001 Aug 7. PMID 11493700
- [Background] Avellino R, Romano S, Parasole R, Bisogni R, Lamberti A, Poggi V, Venuta S, Romano MF. Rapamycin stimulates apoptosis of childhood acute lymphoblastic leukemia cells. Blood. 2005 Aug 15;106(4):1400-6. doi: 10.1182/blood-2005-03-0929. Epub 2005 May 5. PMID 15878982
- [Background] Beuvink I, Boulay A, Fumagalli S, Zilbermann F, Ruetz S, O'Reilly T, Natt F, Hall J, Lane HA, Thomas G. The mTOR inhibitor RAD001 sensitizes tumor cells to DNA-damaged induced apoptosis through inhibition of p21 translation. Cell. 2005 Mar 25;120(6):747-59. doi: 10.1016/j.cell.2004.12.040. PMID 15797377
- [Background] Grunwald V, DeGraffenried L, Russel D, Friedrichs WE, Ray RB, Hidalgo M. Inhibitors of mTOR reverse doxorubicin resistance conferred by PTEN status in prostate cancer cells. Cancer Res. 2002 Nov 1;62(21):6141-5. PMID 12414639
- [Background] Shi Y, Frankel A, Radvanyi LG, Penn LZ, Miller RG, Mills GB. Rapamycin enhances apoptosis and increases sensitivity to cisplatin in vitro. Cancer Res. 1995 May 1;55(9):1982-8. PMID 7728769
- [Background] Xu Q, Thompson JE, Carroll M. mTOR regulates cell survival after etoposide treatment in primary AML cells. Blood. 2005 Dec 15;106(13):4261-8. doi: 10.1182/blood-2004-11-4468. Epub 2005 Sep 8. PMID 16150937
- [Background] Castro AF, Rebhun JF, Clark GJ, Quilliam LA. Rheb binds tuberous sclerosis complex 2 (TSC2) and promotes S6 kinase activation in a rapamycin- and farnesylation-dependent manner. J Biol Chem. 2003 Aug 29;278(35):32493-6. doi: 10.1074/jbc.C300226200. Epub 2003 Jul 3. PMID 12842888
- [Background] Long X, Lin Y, Ortiz-Vega S, Yonezawa K, Avruch J. Rheb binds and regulates the mTOR kinase. Curr Biol. 2005 Apr 26;15(8):702-13. doi: 10.1016/j.cub.2005.02.053. PMID 15854902
- [Background] Kay JE, Kromwel L, Doe SE, Denyer M. Inhibition of T and B lymphocyte proliferation by rapamycin. Immunology. 1991 Apr;72(4):544-9. PMID 1709916
- [Background] Morris RE. Rapamycin: FK506's fraternal twin or distant cousin? Immunol Today. 1991 May;12(5):137-40. doi: 10.1016/S0167-5699(05)80040-4. PMID 1715165
- [Background] Brown VI, Fang J, Alcorn K, Barr R, Kim JM, Wasserman R, Grupp SA. Rapamycin is active against B-precursor leukemia in vitro and in vivo, an effect that is modulated by IL-7-mediated signaling. Proc Natl Acad Sci U S A. 2003 Dec 9;100(25):15113-8. doi: 10.1073/pnas.2436348100. Epub 2003 Dec 1. PMID 14657335
- [Background] Gottschalk AR, Boise LH, Thompson CB, Quintans J. Identification of immunosuppressant-induced apoptosis in a murine B-cell line and its prevention by bcl-x but not bcl-2. Proc Natl Acad Sci U S A. 1994 Jul 19;91(15):7350-4. doi: 10.1073/pnas.91.15.7350. PMID 7518929
- [Background] Hultsch T, Martin R, Hohman RJ. The effect of the immunophilin ligands rapamycin and FK506 on proliferation of mast cells and other hematopoietic cell lines. Mol Biol Cell. 1992 Sep;3(9):981-7. doi: 10.1091/mbc.3.9.981. PMID 1384815
- [Background] Majewski M, Korecka M, Kossev P, Li S, Goldman J, Moore J, Silberstein LE, Nowell PC, Schuler W, Shaw LM, Wasik MA. The immunosuppressive macrolide RAD inhibits growth of human Epstein-Barr virus-transformed B lymphocytes in vitro and in vivo: A potential approach to prevention and treatment of posttransplant lymphoproliferative disorders. Proc Natl Acad Sci U S A. 2000 Apr 11;97(8):4285-90. doi: 10.1073/pnas.080068597. PMID 10759564
- [Background] Muthukkumar S, Ramesh TM, Bondada S. Rapamycin, a potent immunosuppressive drug, causes programmed cell death in B lymphoma cells. Transplantation. 1995 Aug 15;60(3):264-70. doi: 10.1097/00007890-199508000-00010. PMID 7544036
- [Background] Yamamoto-Yamaguchi Y, Okabe-Kado J, Kasukabe T, Honma Y. Induction of differentiation of human myeloid leukemia cells by immunosuppressant macrolides (rapamycin and FK506) and calcium/calmodulin-dependent kinase inhibitors. Exp Hematol. 2001 May;29(5):582-8. doi: 10.1016/s0301-472x(01)00626-9. PMID 11376870
- [Background] Yee KW, Zeng Z, Konopleva M, Verstovsek S, Ravandi F, Ferrajoli A, Thomas D, Wierda W, Apostolidou E, Albitar M, O'Brien S, Andreeff M, Giles FJ. Phase I/II study of the mammalian target of rapamycin inhibitor everolimus (RAD001) in patients with relapsed or refractory hematologic malignancies. Clin Cancer Res. 2006 Sep 1;12(17):5165-73. doi: 10.1158/1078-0432.CCR-06-0764. PMID 16951235
- [Background] Zeng Z, Sarbassov dos D, Samudio IJ, Yee KW, Munsell MF, Ellen Jackson C, Giles FJ, Sabatini DM, Andreeff M, Konopleva M. Rapamycin derivatives reduce mTORC2 signaling and inhibit AKT activation in AML. Blood. 2007 Apr 15;109(8):3509-12. doi: 10.1182/blood-2006-06-030833. Epub 2006 Dec 19. PMID 17179228
- [Background] Eng CP, Sehgal SN, Vezina C. Activity of rapamycin (AY-22,989) against transplanted tumors. J Antibiot (Tokyo). 1984 Oct;37(10):1231-7. doi: 10.7164/antibiotics.37.1231. PMID 6501094
- [Background] Hudes G, Carducci M, Tomczak P, Dutcher J, Figlin R, Kapoor A, Staroslawska E, Sosman J, McDermott D, Bodrogi I, Kovacevic Z, Lesovoy V, Schmidt-Wolf IG, Barbarash O, Gokmen E, O'Toole T, Lustgarten S, Moore L, Motzer RJ; Global ARCC Trial. Temsirolimus, interferon alfa, or both for advanced renal-cell carcinoma. N Engl J Med. 2007 May 31;356(22):2271-81. doi: 10.1056/NEJMoa066838. PMID 17538086
- [Background] Ansell SM, Inwards DJ, Rowland KM Jr, Flynn PJ, Morton RF, Moore DF Jr, Kaufmann SH, Ghobrial I, Kurtin PJ, Maurer M, Allmer C, Witzig TE. Low-dose, single-agent temsirolimus for relapsed mantle cell lymphoma: a phase 2 trial in the North Central Cancer Treatment Group. Cancer. 2008 Aug 1;113(3):508-14. doi: 10.1002/cncr.23580. PMID 18543327
- [Background] Rizzieri DA, Feldman E, Dipersio JF, Gabrail N, Stock W, Strair R, Rivera VM, Albitar M, Bedrosian CL, Giles FJ. A phase 2 clinical trial of deforolimus (AP23573, MK-8669), a novel mammalian target of rapamycin inhibitor, in patients with relapsed or refractory hematologic malignancies. Clin Cancer Res. 2008 May 1;14(9):2756-62. doi: 10.1158/1078-0432.CCR-07-1372. PMID 18451242
- [Background] Chiarini F, Grimaldi C, Ricci F, et al. Temsirolimus, An Allosteric mTORC1 Inhibitor, Is Synergistic with Clofarabine in AML and AML Leukemia Initiating Cells. ASH Annual Meeting Abstracts;118:2596-.
- [Background] Dan S, Naito M, Tsuruo T. Selective induction of apoptosis in Philadelphia chromosome-positive chronic myelogenous leukemia cells by an inhibitor of BCR - ABL tyrosine kinase, CGP 57148. Cell Death Differ. 1998 Aug;5(8):710-5. doi: 10.1038/sj.cdd.4400400. PMID 10200527
- [Background] Duran I, Kortmansky J, Singh D, Hirte H, Kocha W, Goss G, Le L, Oza A, Nicklee T, Ho J, Birle D, Pond GR, Arboine D, Dancey J, Aviel-Ronen S, Tsao MS, Hedley D, Siu LL. A phase II clinical and pharmacodynamic study of temsirolimus in advanced neuroendocrine carcinomas. Br J Cancer. 2006 Nov 6;95(9):1148-54. doi: 10.1038/sj.bjc.6603419. Epub 2006 Oct 10. PMID 17031397
- [Background] Tabernero J, Rojo F, Calvo E, Burris H, Judson I, Hazell K, Martinelli E, Ramon y Cajal S, Jones S, Vidal L, Shand N, Macarulla T, Ramos FJ, Dimitrijevic S, Zoellner U, Tang P, Stumm M, Lane HA, Lebwohl D, Baselga J. Dose- and schedule-dependent inhibition of the mammalian target of rapamycin pathway with everolimus: a phase I tumor pharmacodynamic study in patients with advanced solid tumors. J Clin Oncol. 2008 Apr 1;26(10):1603-10. doi: 10.1200/JCO.2007.14.5482. Epub 2008 Mar 10. PMID 18332469
- [Background] Recher C, Beyne-Rauzy O, Demur C, Chicanne G, Dos Santos C, Mas VM, Benzaquen D, Laurent G, Huguet F, Payrastre B. Antileukemic activity of rapamycin in acute myeloid leukemia. Blood. 2005 Mar 15;105(6):2527-34. doi: 10.1182/blood-2004-06-2494. Epub 2004 Nov 18. PMID 15550488
- [Background] Greenberg PL, Lee SJ, Advani R, Tallman MS, Sikic BI, Letendre L, Dugan K, Lum B, Chin DL, Dewald G, Paietta E, Bennett JM, Rowe JM. Mitoxantrone, etoposide, and cytarabine with or without valspodar in patients with relapsed or refractory acute myeloid leukemia and high-risk myelodysplastic syndrome: a phase III trial (E2995). J Clin Oncol. 2004 Mar 15;22(6):1078-86. doi: 10.1200/JCO.2004.07.048. PMID 15020609
- [Background] Park S, Chapuis N, Marcoux FS, et al. RAD001: A Clinico-Biological Phase I GOELAMS trial of Everolimus Association with High Dose Chemotherapy in Late Relapsing AML Patients Under 65 Years of Age. ASH Annual Meeting Abstracts;118:945-.
- [Background] Barnes JA, Jacobsen E, Feng Y, Freedman A, Hochberg EP, LaCasce AS, Armand P, Joyce R, Sohani AR, Rodig SJ, Neuberg D, Fisher DC, Abramson JS. Everolimus in combination with rituximab induces complete responses in heavily pretreated diffuse large B-cell lymphoma. Haematologica. 2013 Apr;98(4):615-9. doi: 10.3324/haematol.2012.075184. Epub 2012 Nov 9. PMID 23144193
- [Background] Craig FE, Foon KA. Flow cytometric immunophenotyping for hematologic neoplasms. Blood. 2008 Apr 15;111(8):3941-67. doi: 10.1182/blood-2007-11-120535. Epub 2008 Jan 15. PMID 18198345
- [Background] Jennings CD, Foon KA. Recent advances in flow cytometry: application to the diagnosis of hematologic malignancy. Blood. 1997 Oct 15;90(8):2863-92. No abstract available. PMID 9376567
- [Background] Irish JM, Hovland R, Krutzik PO, Perez OD, Bruserud O, Gjertsen BT, Nolan GP. Single cell profiling of potentiated phospho-protein networks in cancer cells. Cell. 2004 Jul 23;118(2):217-28. doi: 10.1016/j.cell.2004.06.028. PMID 15260991
- [Background] Jacobberger JW, Sramkoski RM, Frisa PS, Ye PP, Gottlieb MA, Hedley DW, Shankey TV, Smith BL, Paniagua M, Goolsby CL. Immunoreactivity of Stat5 phosphorylated on tyrosine as a cell-based measure of Bcr/Abl kinase activity. Cytometry A. 2003 Aug;54(2):75-88. doi: 10.1002/cyto.a.10063. PMID 12879454
- [Background] Perez OD, Nolan GP. Simultaneous measurement of multiple active kinase states using polychromatic flow cytometry. Nat Biotechnol. 2002 Feb;20(2):155-62. doi: 10.1038/nbt0202-155. PMID 11821861
- [Background] Krutzik PO, Irish JM, Nolan GP, Perez OD. Analysis of protein phosphorylation and cellular signaling events by flow cytometry: techniques and clinical applications. Clin Immunol. 2004 Mar;110(3):206-21. doi: 10.1016/j.clim.2003.11.009. PMID 15047199
- [Background] Chow S, Hedley D, Grom P, Magari R, Jacobberger JW, Shankey TV. Whole blood fixation and permeabilization protocol with red blood cell lysis for flow cytometry of intracellular phosphorylated epitopes in leukocyte subpopulations. Cytometry A. 2005 Sep;67(1):4-17. doi: 10.1002/cyto.a.20167. PMID 16080188
- [Background] Chow S, Minden MD, Hedley DW. Constitutive phosphorylation of the S6 ribosomal protein via mTOR and ERK signaling in the peripheral blasts of acute leukemia patients. Exp Hematol. 2006 Sep;34(9):1183-91. doi: 10.1016/j.exphem.2006.05.002. PMID 16939811
- [Background] Hedley DW, Chow S, Goolsby C, Shankey TV. Pharmacodynamic monitoring of molecular-targeted agents in the peripheral blood of leukemia patients using flow cytometry. Toxicol Pathol. 2008 Jan;36(1):133-9. doi: 10.1177/0192623307310952. PMID 18337231
- [Background] Tong FK, Chow S, Hedley D. Pharmacodynamic monitoring of BAY 43-9006 (Sorafenib) in phase I clinical trials involving solid tumor and AML/MDS patients, using flow cytometry to monitor activation of the ERK pathway in peripheral blood cells. Cytometry B Clin Cytom. 2006 May;70(3):107-14. doi: 10.1002/cyto.b.20092. PMID 16498671
- [Background] Vignot S, Faivre S, Aguirre D, Raymond E. mTOR-targeted therapy of cancer with rapamycin derivatives. Ann Oncol. 2005 Apr;16(4):525-37. doi: 10.1093/annonc/mdi113. Epub 2005 Feb 22. PMID 15728109
- [Background] Chan S. Targeting the mammalian target of rapamycin (mTOR): a new approach to treating cancer. Br J Cancer. 2004 Oct 18;91(8):1420-4. doi: 10.1038/sj.bjc.6602162. PMID 15365568
- [Background] Punt CJ, Boni J, Bruntsch U, Peters M, Thielert C. Phase I and pharmacokinetic study of CCI-779, a novel cytostatic cell-cycle inhibitor, in combination with 5-fluorouracil and leucovorin in patients with advanced solid tumors. Ann Oncol. 2003 Jun;14(6):931-7. doi: 10.1093/annonc/mdg248. PMID 12796032
- [Background] Witzig TE, Geyer SM, Ghobrial I, Inwards DJ, Fonseca R, Kurtin P, Ansell SM, Luyun R, Flynn PJ, Morton RF, Dakhil SR, Gross H, Kaufmann SH. Phase II trial of single-agent temsirolimus (CCI-779) for relapsed mantle cell lymphoma. J Clin Oncol. 2005 Aug 10;23(23):5347-56. doi: 10.1200/JCO.2005.13.466. Epub 2005 Jun 27. PMID 15983389
- [Background] Scott EC, Perl A, Luger SM, Carroll M, Kasner M. A Feasibility Study of Rapamycin with Hyper-CVAD Chemotherapy in Adults with Acute Lymphoblastic Leukemia (ALL) and Other Aggressive Lymphoid Malignancies and Evaluation of mTOR Signaling Using Phosphoflow. ASH Annual Meeting Abstracts;118:4245-.
- [Background] Keijzer A, van der Valk P, Ossenkoppele GJ, van de Loosdrecht AA. Mucormycosis in a patient with low risk myelodysplasia treated with anti-TNF-alpha. Haematologica. 2006 Dec;91(12 Suppl):ECR51. PMID 17194657
- [Background] Vasquez EM. Sirolimus: a new agent for prevention of renal allograft rejection. Am J Health Syst Pharm. 2000 Mar 1;57(5):437-48; quiz 449-51. doi: 10.1093/ajhp/57.5.437. PMID 10711524
- [Background] Berman E, Heller G, Santorsa J, McKenzie S, Gee T, Kempin S, Gulati S, Andreeff M, Kolitz J, Gabrilove J, et al. Results of a randomized trial comparing idarubicin and cytosine arabinoside with daunorubicin and cytosine arabinoside in adult patients with newly diagnosed acute myelogenous leukemia. Blood. 1991 Apr 15;77(8):1666-74. PMID 2015395
- [Background] Robert J. Clinical pharmacokinetics of idarubicin. Clin Pharmacokinet. 1993 Apr;24(4):275-88. doi: 10.2165/00003088-199324040-00002. PMID 8491056
- [Background] Berman E. A review of idarubicin in acute leukemia. Oncology (Williston Park). 1993 Oct;7(10):91-8, 104; discussion 104-7. PMID 8251309
- [Background] Buckley MM, Lamb HM. Oral idarubicin. A review of its pharmacological properties and clinical efficacy in the treatment of haematological malignancies and advanced breast cancer. Drugs Aging. 1997 Jul;11(1):61-86. doi: 10.2165/00002512-199711010-00006. PMID 9237041
- [Background] Hollingshead LM, Faulds D. Idarubicin. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential in the chemotherapy of cancer. Drugs. 1991 Oct;42(4):690-719. doi: 10.2165/00003495-199142040-00010. PMID 1723369
- [Background] Hines JD, Oken MM, Mazza JJ, Keller AM, Streeter RR, Glick JH. High-dose cytosine arabinoside and m-AMSA is effective therapy in relapsed acute nonlymphocytic leukemia. J Clin Oncol. 1984 Jun;2(6):545-9. doi: 10.1200/JCO.1984.2.6.545. PMID 6233399
- [Background] Early AP, Preisler HD, Slocum H, Rustum YM. A pilot study of high-dose 1-beta-D-arabinofuranosylcytosine for acute leukemia and refractory lymphoma: clinical response and pharmacology. Cancer Res. 1982 Apr;42(4):1587-94. PMID 6949642
- [Background] Salinsky MC, Levine RL, Aubuchon JP, Schutta HS. Acute cerebellar dysfunction with high-dose ARA-C therapy. Cancer. 1983 Feb 1;51(3):426-9. doi: 10.1002/1097-0142(19830201)51:33.0.co;2-s. PMID 6571798
- [Background] Lass JH, Lazarus HM, Reed MD, Herzig RH. Topical corticosteroid therapy for corneal toxicity from systemically administered cytarabine. Am J Ophthalmol. 1982 Nov;94(5):617-21. doi: 10.1016/0002-9394(82)90006-x. PMID 6756155
- [Background] Nand S, Messmore HL Jr, Patel R, Fisher SG, Fisher RI. Neurotoxicity associated with systemic high-dose cytosine arabinoside. J Clin Oncol. 1986 Apr;4(4):571-5. doi: 10.1200/JCO.1986.4.4.571. PMID 3457102
- [Background] Herzig RH, Herzig GP, Wolff SN, Hines JD, Fay JW, Phillips GL. Central nervous system effects of high-dose cytosine arabinoside. Semin Oncol. 1987 Jun;14(2 Suppl 1):21-4. No abstract available. PMID 3589694
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org